CLINICAL TRIAL: NCT07243899
Title: The Multimodal Model Predicts the Efficacy of Immunotherapy Checkpoint Inhibitors Combined With Chemotherapy for the Treatment of Advanced Non-small Cell Lung Cancer and the Occurrence Risk of Chemotherapy-induced Pneumonitis
Brief Title: Multimodal Model Predicts Treatment Efficacy and CIP Risk in Advanced NSCLC With Immunotherapy and Chemotherapy
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2025-594R
Record Dates: First submitted 2025-11-15; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort: for feature selection and model construction
  Interventions: Other: This study is an observational study; the intervention is not applicable.
- Internal validation cohort: for hyperparameter optimization and overfitting monitoring
  Interventions: Other: This study is an observational study; the intervention is not applicable.
- External validation cohort: an independent cohort for final model validation
  Interventions: Other: This study is an observational study; the intervention is not applicable.

INTERVENTIONS:
Other: This study is an observational study; the intervention is not applicable. — This study is an observational study; the intervention is not applicable.

SUMMARY:
Immunotherapy is a crucial first-line treatment for advanced non-small cell lung cancer (NSCLC) without gene mutations. However, chemotherapy-induced pneumonitis (CIP) is a common adverse effect of immunotherapy, with severe cases even posing a threat to life. Therefore, identifying effective biomarkers and models for predicting the efficacy of immunotherapy in NSCLC is of great significance. At present, there is still a lack of effective predictive indicators in clinical practice. This study aims to construct a multimodal model based on factors such as chest CT, pulmonary function, cellular immunity, and cytokine levels to accurately predict the efficacy of combined therapy and the occurrence of related adverse reactions in NSCLC, in order to provide a reference for individualized treatment.

DETAILED DESCRIPTION:
This is an observational cross-sectional retrospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Consistent with the "Chinese Medical Association Guidelines for the Diagnosis and Treatment of Lung Cancer (2018 Edition)," histologically confirmed as NSCLC;
2. According to the 8th edition of the AJCC TNM staging system, it is stage III B to IV and not suitable for surgery;
3. Age ≥18 years;
4. First-time recipients of immunotherapy combined with chemotherapy;
5. Baseline data within 1 month before the start of treatment is complete (at least including chest CT, pulmonary function, and laboratory tests);
6. At least 1 measurable lesion according to RECIST 1.1;
7. Receiving immune checkpoint inhibitor therapy for more than 2 cycles;
8. Clinical data is complete.

Exclusion Criteria:

1. Presence of other malignant tumors;
2. Previous exposure to immunotherapy or systemic chemotherapy;
3. Patients with severe dysfunction of vital organs (heart, liver, lungs, kidneys) and bone marrow at baseline;
4. Presence of severe infectious diseases, active autoimmune diseases, or immune deficiencies that significantly affect immune function;
5. Organ transplantation;
6. Pregnant or lactating women;
7. Incomplete clinical treatment or follow-up information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with inoperable stage IIIB to IV NSCLS using immune checkpoint inhibitors in combination with chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From first dose through 31 August 2025, corresponding to a maximum follow-up of approximately 5.5 years (~290 weeks).
  Time from the first dose of immune-checkpoint inhibitor plus chemotherapy to the earliest date of radiologic progression (per RECIST 1.1) or death from any cause.

SECONDARY OUTCOMES:
The disease control rate (DCR) | Tumor response assessed every 6 weeks (±1 week) for up to 24 weeks or until progression/death/cut-off (31 Aug 2025); the proportion will be calculated from the best response recorded within the first 24 weeks (4 cycles) per RECIST 1.1.
  Proportion of patients achieving complete response (CR), partial response (PR), or stable disease (SD) as best overall response per RECIST 1.1.
Checkpoint inhibitor pneumonitis (CIP) | Within 4 months after the initiation of immunotherapy combined with chemotherapy.
  an immune-related adverse event (irAE) endpoint refers to new pulmonary infiltrates on chest imaging after immune checkpoint inhibitor (ICI) treatment, accompanied by dyspnea and/or other respiratory signs/symptoms (including cough and exertional dyspnea), excluding new pulmonary infections or tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Nuo Xu, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No